CLINICAL TRIAL: NCT00177008
Title: Aripiprazole for the Treatment of Schizophrenia With Co-Morbid Social Anxiety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4680
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2007-01-29 (Estimated); Status verified 2007-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Social Anxiety Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Social Anxiety Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Phobia, Social | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
This study will determine the efficacy of a medication switch to Aripiprazole for the treatment of schizophrenia or schizoaffective disorder in patients with moderate to high symptoms of social anxiety. Specifically the study will test the possibility that a medication switch to Aripiprazole reduces symptoms of social anxiety in this patient population.

DETAILED DESCRIPTION:
Although research has shown that social anxiety is very common among patients suffering from schizophrenia or schizoaffective disorder, it is rarely diagnosed and treated in this patient population. This study will determine the efficacy of a medication switch to Aripiprazole for the treatment of schizophrenia in patients with moderate to high symptoms of social anxiety. Specifically the study will test the possibility that a medication switch to Aripiprazole reduces symptoms of social anxiety in this patient population. In addition, the study will test the possibility that Aripiprazole significantly improves social adjustment, quality of life and level of functioning in these patients. The study may also assess the ability of Aripiprazole to reduce sexual dysfunction.

ELIGIBILITY:
Inclusion Criteria

1. Patients meeting DSM IV diagnostic criteria for schizophrenia or schizoaffective disorder.
2. Patients presenting with comorbid social anxiety symptoms of moderate to high severity are eligible for participation in the study. Only patients with LSAS scores above 30* qualify for the study.
3. Age 18-65
4. Gender: males or females
5. Females: non-pregnant, not of child-bearing potential; if of child-bearing age must be on contraceptive such as pill or shot (condom alone not sufficient)
6. Good general health

Exclusion Criteria:

1. Patient does not meet DSM IV diagnostic criteria for schizophrenia or schizoaffective disorder
2. Patient carries a diagnosis of dementia, degenerative CNS disorders, mental retardation, substance abuse or dependence other than nicotine dependence or alcohol abuse will be excluded from the study.
3. Patients with acute medical conditions are not eligible.
4. Patients allergic or otherwise intolerant or non-responsive to Aripiprazole
5. Patient with history of suicidal, homicidal or assaultive plans or attempts in the past 6 months.
6. Clinically significant EKG or lab abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2004-03; Study Completion 2007-01

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale- Change from Baseline to Final Visit
Sheehan Disability Scale- Change from Baseline to Final Visit
Lehman Quality of Life Interview- Change from Baseline to Final Visit

SECONDARY OUTCOMES:
Instrumental Activities of Daily Living-Change from Baseline to Final Visit
Clinical Global Impression scales [CGI]and [CGI-C]- change from Baseline to Final Visit.
Ultimate game paradigm as a measure of social cohesion- Change from Baseline to Final Visit
Arizona sexual dysfunction scale- Change from Baseline to Final Visit
COSAPSQ -Change from Baseline to Final Visit
HAM-D-Change from Baseline to Final Visit
PANSS- Change from Baseline to Final Visit
CAGE -Change from Baseline to Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Petti, MD, MPH, Principal Investigator — Rutgers, The State University of New Jersey; Robert Stern, MD, Study Director — UMDNJ-RWJMS
Locations (1):
- Robert Wood Johnson Medical School - Psychiatry Dept., Piscataway, New Jersey, United States

REFERENCES:
- [Background] Kendler KS, Gallagher TJ, Abelson JM, Kessler RC. Lifetime prevalence, demographic risk factors, and diagnostic validity of nonaffective psychosis as assessed in a US community sample. The National Comorbidity Survey. Arch Gen Psychiatry. 1996 Nov;53(11):1022-31. doi: 10.1001/archpsyc.1996.01830110060007. PMID 8911225
- [Background] Cassano GB, Pini S, Saettoni M, Rucci P, Dell'Osso L. Occurrence and clinical correlates of psychiatric comorbidity in patients with psychotic disorders. J Clin Psychiatry. 1998 Feb;59(2):60-8. doi: 10.4088/jcp.v59n0204. PMID 9501887
- [Background] Cosoff SJ, Hafner RJ. The prevalence of comorbid anxiety in schizophrenia, schizoaffective disorder and bipolar disorder. Aust N Z J Psychiatry. 1998 Feb;32(1):67-72. doi: 10.3109/00048679809062708. PMID 9565185
- [Background] Penn DL, Hope DA, Spaulding W, Kucera J. Social anxiety in schizophrenia. Schizophr Res. 1994 Feb;11(3):277-84. doi: 10.1016/0920-9964(94)90022-1. PMID 8193064
- [Background] Blanchard JJ, Mueser KT, Bellack AS. Anhedonia, positive and negative affect, and social functioning in schizophrenia. Schizophr Bull. 1998;24(3):413-24. doi: 10.1093/oxfordjournals.schbul.a033336. PMID 9718633
- [Background] Liebowitz MR. Social phobia. Mod Probl Pharmacopsychiatry. 1987;22:141-73. doi: 10.1159/000414022. No abstract available. PMID 2885745
- [Background] Bobes J. How is recovery from social anxiety disorder defined? J Clin Psychiatry. 1998;59 Suppl 17:12-9. PMID 9811425
- [Background] Stern RG, Frank D, Meraj H, Ballou S, Schnur E,: High social phobia scale scores in schizophrenia do not correlate with psychosis symptom severity scores. New Research Program and Abstracts. American Psychiatric Association 151st Annual Meeting, Washington, D.C, May 1999, NR 239.
- [Background] Lehman AF, Ward NC, Linn LS. Chronic mental patients: the quality of life issue. Am J Psychiatry. 1982 Oct;139(10):1271-6. doi: 10.1176/ajp.139.10.1271. PMID 7124978
- [Background] Stern RG, Frank D, Farooq S, Beyer M,: The relationship of social anxiety to level of function over time in patients with schizophrenia. Presented at the 2002 Annual Meeting of the APA, Philadelphia, Pa.
- [Background] Stern RG, Frank D, Farooq S, Beyer M: Social anxiety symptoms are common severe and unrelated to psychosis - A replication study. New Research Program and Abstracts. American Psychiatric Association 2002, Philadelphia, Pa.
- [Background] Jordan S, Koprivica V, Chen R, Tottori K, Kikuchi T, Altar CA. The antipsychotic aripiprazole is a potent, partial agonist at the human 5-HT1A receptor. Eur J Pharmacol. 2002 Apr 26;441(3):137-40. doi: 10.1016/s0014-2999(02)01532-7. PMID 12063084
- [Background] Sramek JJ, Zarotsky V, Cutler NR. Generalised anxiety disorder: treatment options. Drugs. 2002;62(11):1635-48. doi: 10.2165/00003495-200262110-00005. PMID 12109925
- [Background] Leslie RA. Gepirone. Organon. Curr Opin Investig Drugs. 2001 Aug;2(8):1120-7. PMID 11892924
- [Background] Bourin M, Hascoet M. Drug mechanisms in anxiety. Curr Opin Investig Drugs. 2001 Feb;2(2):259-65. PMID 11816841
- [Background] Mennin DS, Fresco DM, Heimberg RG, Schneier FR, Davies SO, Liebowitz MR. Screening for social anxiety disorder in the clinical setting: using the Liebowitz Social Anxiety Scale. J Anxiety Disord. 2002;16(6):661-73. doi: 10.1016/s0887-6185(02)00134-2. PMID 12405524